CLINICAL TRIAL: NCT04333121
Title: Modelling Predictive gender-and Gestation-specific Weight Reference Centiles for Preterm Infants Using a Population-based Cohort Study at Neonatology Unit of Assuit University Children Hospital
Brief Title: Modelling Weight Reference Centiles for Preterm Infants
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khalaf Ali, Modelling predictive gender-and gestation-specific weight reference centiles for preterm infants using a population-based cohort study at neonatology unit of Assuit University Children Hospital, Assiut University
Other Study IDs: weight chart for preterms
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Pre-Term
MeSH Terms: conditions — Premature Birth | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: weight — we can monitoring the growth of the infants by weight gain degree

SUMMARY:
The aim of this study is to model longitudinal data at NICU of Assuit University Children Hospital to create predictive growth charts for weight in preterm infants from birth till discharge, that take into account the differing growth rates post-birth when compared to in-utero growth ,and to compare it with WHO chart for preterms.

DETAILED DESCRIPTION:
It is an observational retrospective study achieved by collecting retrospective, longitudinal measurements of weight from preterm infants born at <34 weeks gestation, starting from birth, and model gender- and gestation specific predictive centile charts till discharge from the neonatal unit by a population-based cohort study.

ELIGIBILITY:
Inclusion Criteria:

* Data will be collected for all infants born at <34 weeks of gestation who were delivered by vaginal or caesarian section and born at Assuit University Hospital or referred to it.

Exclusion Criteria:

* (1) Any neonate born at 34 weeks of gestation or more, (2) any neonate born at <34 weeks of gestation who died before a second weight could be recorded.

Ages: 1 Day to 1 Month | Sex: All
Age Groups: Child
Gender Based: Yes — we will compare the difference of weight gain between males and females infants
Study Population: It is an observational retrospective study achieved by collecting retrospective, longitudinal measurements of weight from preterm infants born at <34 weeks gestation, starting from birth, and model gender- and gestation specific predictive centile charts till discharge from the neonatal unit by a population-based cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Modelling predictive gender-and gestation-specific weight reference centiles for preterm infants using a population-based cohort study at neonatology unit of Assuit University Children Hospital | one year
  It is an observational retrospective study achieved by collecting retrospective, longitudinal measurements of weight from preterm infants born at <34 weeks gestation, starting from birth, and model gender- and gestation specific predictive centile charts till discharge from the neonatal unit by a population-based cohort study.

REFERENCES:
- [Background] Dusick AM, Poindexter BB, Ehrenkranz RA, Lemons JA. Growth failure in the preterm infant: can we catch up? Semin Perinatol. 2003 Aug;27(4):302-10. doi: 10.1016/s0146-0005(03)00044-2. PMID 14510321
- [Background] Secher NJ, Kern Hansen P, Thomsen BL, Keiding N. Growth retardation in preterm infants. Br J Obstet Gynaecol. 1987 Feb;94(2):115-20. doi: 10.1111/j.1471-0528.1987.tb02336.x. PMID 3548805